CLINICAL TRIAL: NCT06691672
Title: Feasibility Study of Dialysis Clinic Semi-Autonomous Ultrasound Scanning Using the Vexev Ultrasound Imaging System for Arteriovenous Fistula Mapping Examinations.
Brief Title: Feasibility Study of Dialysis Clinic Semi-Autonomous Ultrasound Scanning Using the Vexev Ultrasound Imaging System for Arteriovenous Fistula Mapping Examinations. The CANSCAN Trial.
Acronym: CANSCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vexev Pty Ltd (Industry)
Collaborators: USRC Kidney Research (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIP-3-20242468
Record Dates: First submitted 2024-11-12; First posted 2024-11-15 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Feasibility Assessment of the VxWave Device for Vascular Access Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imaging Arm (Experimental)
  Interventions: Diagnostic Test: Robotic Tomographic ultrasound imaging of the arm vasculature.

INTERVENTIONS:
Diagnostic Test: Robotic Tomographic ultrasound imaging of the arm vasculature. — Semi-autonomous robotic tomographic ultrasound imaging of the arm vasculature for vascular access creation mapping in CKD patients.

SUMMARY:
Study to assess the feasibility of dialysis clinic staff to perform upper limb mapping ultrasound scans using the Vexev Ultrasound Imaging System.

ELIGIBILITY:
Inclusion Criteria:

1. Referred to a study site for chronic renal replacement therapy OR referred to a study site for management of CKD.
2. Able to understand the procedures and requirements of the study and provide written informed consent and authorization for protected health information disclosure.
3. Greater than or equal to 21 years of age at the time of written informed consent.

Exclusion Criteria:

1. Patients' unable to load arm into scanning bed (due to upper limb medical co-morbidities/injury).
2. Patient has evidence of open or incompletely healed wounds on both arms. Patients with open or incompletely healed wounds on a single arm are not excluded - if the ipsilateral arm is not able to be scanned - contralateral arm may be scanned.
3. Any acute or chronic condition that would limit the ability of the patient to participate in the study - in the opinion of the principal investigator.
4. Previous vascular/vascular access surgery on both upper limbs. Patients with previous vascular/vascular access surgery on a single arm are not excluded- contralateral arm may be scanned.

   -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Vascular Access Robotic Tomographic Ultrasound (RTU) Mapping Efficacy and Feasability | From enrollment to the end of viable assessment window at 90 days.
  The proportion of RTU vascular mapping scans performed using the VxWave Vascular Ultrasound Imaging Device that are assessed by interventionalists to provide sufficient imaging data to determine vascular access options.

CONTACTS AND LOCATIONS:
Locations (1):
- USRC E Houston Street, San Antonio, Texas, United States